CLINICAL TRIAL: NCT05023083
Title: Cross Cultural Adaptation of Functional Status Questionnaire (FSQ) in Urdu Language in CABG Patients
Brief Title: Cross Cultural Adaptation of Functional Status Questionnaire in Urdu Language in CABG Patients
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/20/049 Ghazal Jamshaid
Record Dates: First submitted 2021-05-19; First posted 2021-08-26 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: CABG; Post-cardiac Surgery
Keywords: ADLs; CABG; Functional Status Questionnaire; FSQ; Quality of life.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diseased individuals: post CABG patients will be included in the study to fill the tool
  Interventions: Other: Functional Status Questionnaire Urdu version; Other: Original Functional Status Questionnaire
- healthy individuals: 20 healthy individual will be included to solve questionnaire
  Interventions: Other: Functional Status Questionnaire Urdu version; Other: Original Functional Status Questionnaire

INTERVENTIONS:
Other: Functional Status Questionnaire Urdu version — The FSQ instrument translated into Urdu consists of only 34 items, main sections addressed physical function in the activities of daily living, psychological function, role function, social function and variety of performance measures.(8) Scores range from a 0 - 4, 1 - 4, and 1 - 6 scale per question depending on section. It increases reliability and patients ease and comfort. Total score range from 0 to 100 higher score represents the more severe condition.
  Other Names: FSQ Urdu version; UFSQ
Other: Original Functional Status Questionnaire — FSQ was developed to allow the comprehensive and efficient assessment of physical, psychosocial, social, and role functioning in ambulatory patients. It is a self-administered survey that takes approximately 15 min to complete. The results can be scored to produce a one-page report for clinicians to use in their practices. The responses to items within a scale are averaged and transformed to a scale with a potential range of 0 to 100.Higher score represents the more severe condition.
  Other Names: FSQ

SUMMARY:
Aim of the study is to create an Urdu version of FSQ which will be of great importance for further research in field of cardiopulmonary physiotherapy, specially to make comparison across the population. We therefor aimed to develop a linguistically validated and reliable Urdu version of FSQ.

DETAILED DESCRIPTION:
The Functional Status Questionnaire (FSQ) is a self-administered functional assessment that provides information on the patient's physical, psychological, social and role functions. The Functional Status Questionnaire is easier and more feasible to complete in short duration of time than the long forms. The FSQ was originally developed in English. It has been translated and validated in several languages and showed excellent reliability and responsiveness. The FSQ questionnaire is translated in Urdu to assess general health, ADLs and functional status of Post Coronary artery bypass graft surgery(CABG) patients. Translation will be performed by two independent translators going through all the steps following the guidelines. The two synthesized translations and the two back translations will be merged into one pre- final version of Urdu FSQ. The expert panel will then compare the conceptual equivalence, experiential equivalence, linguistic equivalence and metric equivalence. After this the final version of Urdu FSQ will be evaluated for validity in 50 Post CABG patients after getting their informed consent to participate in the study and their demographic characteristics. Inclusion criteria involves male and female patients of age between 40 to 60 years (ambulatory). Exclusion criteria includes patients with disability that prevent independent walking, acute cardiac condition, neurological conditions, cognitive impaired problem etc. Reliability and validity of FSQ Urdu version will be evaluated. It has been translated and validated in several languages and showed excellent reliability and responsiveness. However up to-date there is no validated Urdu version of the FSQ available. So, it is essential to translate FSQ in Urdu language to make it more comprehensive for local population who doesn't have command on English language. The purpose of this study is cross-cultural translation of the FSQ into Urdu language and to validate it into Urdu speaking population.

Hence, this study is aimed to produce the Urdu version for Urdu speaking countries, it will have a great significance for the physiotherapists, researchers and educators to assess CABG patients general health, QoL, functional status and ADLs where time is short because FSQ makes it easier to collect data from large populations in comparatively lesser time than long assessment forms.

ELIGIBILITY:
Inclusion Criteria:

* Able to read Urdu language
* Participating in community
* Patient is in ambulatory condition
* Post coronary artery bypass graft (CABG) Patients

Exclusion Criteria:

* Acute Cardiac event (e.g. myocardial infarction (MI), arrhythmia, angina) or intervention (e.g. percutaneous coronary intervention (PCI, valve repair, pacemaker fitting)
* Any other disability or neurological condition Cognitive issue Unwilling to participate

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy and 50 post CABG patients are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Translation of Functional Status Questionnaire(FSQ) | 6 months
  Translation of Functional Status Questionnaire(FSQ) into Urdu Language for using this tool in Pakistani Population who understand Urdu.
Validity of Translated Tool | 6 months
  Validity is assessed for checking that the Translation of Functional Status Questionnaire(FSQ) is valid for using in post-CABG patients in Pakistan.
Reliability of Translated Tool | 6 months
  Reliability is assessed for checking that the Translation of Functional Status Questionnaire(FSQ) is reliable for using in post-CABG patients in Pakistan.

OTHER OUTCOMES:
Functional Status Questionnaire (FSQ) | 15 min
  The FSQ assesses physical function: basic activities of daily living (BADL) and intermediate activities of daily living (IADL), Mental function, social or role function, social activity and quality of social interaction. The FSQ also contains six single items which ask questions about work status, days spent in bed due to illness, days where the patient had to curtail his/her routine activities because of illness, satisfaction with sexual activities, frequency of social interaction and a question about overall health satisfaction. There are 34 items in the FSQ in total. Using a simple algorithm, computer-generated scores are obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Mayo hospital Lahore, Lahore, Asia, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Araujo AM, Miguel JA, Gava EC, de Oliveira BH. Translation and cross-cultural adaptation of an instrument designed for the assessment of quality of life in orthognatic patients. Dental Press J Orthod. 2013 Sep-Oct;18(5):99-106. doi: 10.1590/s2176-94512013000500017. PMID 24352395
- [Background] Davide Castagno M, MB BW, Erland Erdmann M, Faiez Zannad M, Remme WJ, Lopez-Sendon JL, et al. Evaluation of the Functional Status Questionnaire in heart. Am J Cardiol. 1996;78:890-5.
- [Background] Helou AS, Ramos AEB, Oliveira ASB, Quadros AAJ, Fávero FM. The use of functionality scales in patients with Post-Polio Syndrome. Brazilian Journal of Biological Sciences. 2019;6(13):367-79
- [Background] Cleary PD, Jette AM. Reliability and validity of the Functional Status Questionnaire. Quality of Life Research. 2000;9(1):747-53.
- [Background] Einarsson G, Grimby G. Disability and handicap in late poliomyelitis. Scand J Rehabil Med. 1990;22(2):113-21. PMID 2363025
- [Background] Baker GA, Gagnon D, McNulty P. The relationship between seizure frequency, seizure type and quality of life: findings from three European countries. Epilepsy Res. 1998 May;30(3):231-40. doi: 10.1016/s0920-1211(98)00010-2. PMID 9657650
- [Background] van Hout B, Gagnon D, Souetre E, Ried S, Remy C, Baker G, Genton P, Vespignani H, McNulty P. Relationship between seizure frequency and costs and quality of life of outpatients with partial epilepsy in France, Germany, and the United Kingdom. Epilepsia. 1997 Nov;38(11):1221-6. doi: 10.1111/j.1528-1157.1997.tb01220.x. PMID 9579924
- [Background] Jette AM, Davies AR, Cleary PD, Calkins DR, Rubenstein LV, Fink A, Kosecoff J, Young RT, Brook RH, Delbanco TL. The Functional Status Questionnaire: reliability and validity when used in primary care. J Gen Intern Med. 1986 May-Jun;1(3):143-9. doi: 10.1007/BF02602324. PMID 3772582
- [Background] Febriana D, Juanita J, Nurhasanah N. Psychometric Evaluation of Instruments Measuring The Older Adult's Functional Status in Indonesian. Jurnal Keperawatan Padjadjaran. 2019;7(2)
- [Background] Akosile CO, Mgbeojedo UG, Maruf FA, Okoye EC, Umeonwuka IC, Ogunniyi A. Depression, functional disability and quality of life among Nigerian older adults: Prevalences and relationships. Arch Gerontol Geriatr. 2018 Jan;74:39-43. doi: 10.1016/j.archger.2017.08.011. Epub 2017 Sep 6. PMID 28954240
- [Background] Gallanagh S, Castagno D, Wilson B, Erdmann E, Zannad F, Remme WJ, Lopez-Sendon JL, Lechat P, Follath F, Hoglund C, Mareev V, Sadowski Z, Seabra-Gomes RJ, Dargie HJ, McMurray JJ. Evaluation of the functional status questionnaire in heart failure: a sub-study of the second cardiac insufficiency bisoprolol survival study (CIBIS-II). Cardiovasc Drugs Ther. 2011 Feb;25(1):77-85. doi: 10.1007/s10557-011-6284-x. PMID 21287410
- [Background] Swan BA, Maislin G, Traber KB. Symptom distress and functional status changes during the first seven days after ambulatory surgery. Anesth Analg. 1998 Apr;86(4):739-45. doi: 10.1097/00000539-199804000-00012. PMID 9539594
- [Background] Murphy N, Confavreux C, Haas J, Konig N, Roullet E, Sailer M, Swash M, Young C, Merot JL. Quality of life in multiple sclerosis in France, Germany, and the United Kingdom. Cost of Multiple Sclerosis Study Group. J Neurol Neurosurg Psychiatry. 1998 Oct;65(4):460-6. doi: 10.1136/jnnp.65.4.460. PMID 9771766
- [Background] Tedesco C, Manning S, Lindsay R, Alexander C, Owen R, Smucker ML. Functional assessment of elderly patients after percutaneous aortic balloon valvuloplasty: New York Heart Association classification versus functional status questionnaire. Heart Lung. 1990 Mar;19(2):118-25. PMID 2318655